CLINICAL TRIAL: NCT00933829
Title: Comparison of Cosmetic Outcomes of Lacerations of the Trunk and Extremity Repaired Using Absorbable Versus Non-absorbable Sutures
Brief Title: Comparison of Cosmetic Outcomes of Lacerations Repaired Using Absorbable Versus Non-absorbable Sutures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12177
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Lacerations; Wounds; Injuries
Keywords: absorbable sutures; non-absorbable sutures; wound management
MeSH Terms: conditions — Lacerations; Wounds and Injuries | interventions — Sutures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-absorbable arm (Placebo Comparator): uses non-absorbable suture such as Prolene to repair lacerations
  Interventions: Device: Non-absorbable suture (Prolene); Procedure: suture
- Absorbable Suture Arm (Active Comparator): uses absorbable sutures to repair lacerations
  Interventions: Procedure: Absorbable Suture Arm; Procedure: suture

INTERVENTIONS:
Procedure: Absorbable Suture Arm — use of irradiated polyglactin 910
  Other Names: Vicryl Rapide
  Arms: Absorbable Suture Arm
Device: Non-absorbable suture (Prolene) — suture
  Arms: Non-absorbable arm
Procedure: suture — non-absorable sutures and absorable sutures

SUMMARY:
The primary objective of this prospective, randomized study is to compare cosmetic outcomes between absorbable and non-absorbable sutures in truncal and extremity lacerations in the pediatric and adult population. Secondary outcome measures include wound complications such as infection and wound dehiscence at the initial visit; and parental satisfaction and keloid formation after three months post repair.

DETAILED DESCRIPTION:
Even though there some studies showing good outcomes using absorbable sutures in skin closure in clean surgical wounds, ED based studies still need to be conducted to convince ED physicians that the use of absorbable sutures to close the skin in traumatic lacerations are just as acceptable as traditional non-absorbable sutures. Use of absorbable sutures confers several advantages over non-absorbable sutures. For one, patients do not need an additional physician visit either in the office, or more often that not, in the emergency department. These visits add to ED overcrowding, prolonged length of ED stay and are often not reimbursed if seen in the emergency department. Moreover, adult patients need to miss work or school and children often have to miss school or daycare to have these sutures removed. The potential to avert another traumatic experience from suture removal in children who had been restrained for suture placement is another advantage of using absorbable sutures over non-absorbable sutures.

ELIGIBILITY:
Inclusion Criteria:

1. Isolated injury
2. Non-contaminated or minimally contaminated wounds
3. Linear laceration 1-5 cms
4. Topical adhesives not indicated

Exclusion Criteria:

1. Trunk and extremity lacerations less than 1 cm or greater than 5 cm.
2. Moderately contaminated wounds or dirty wounds
3. Wounds with visible foreign bodies
4. Wounds more than 8 hours old
5. Wounds that can be repaired using topical adhesives
6. Complex wounds needing surgical referral
7. Wounds caused by mammalian bites
8. Wounds in patients with immune deficiency, pregnancy, diabetes, suspected bleeding disorder or renal dysfunction
9. Wounds in patients who are currently taking steroids
10. Wounds in areas of tension such as the joint or crease
11. Patients with allergic reaction to the topical anesthetic
12. Irregular wounds

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome is cosmetic outcomes at 3 to 4 months using the visual analogue scale. | at least 3 months post-injury

SECONDARY OUTCOMES:
Secondary outcome measures: complication rates such as infection and dehiscence rates at the first visit post-injury. | 8-12 days post-injury

CONTACTS AND LOCATIONS:
Overall Officials: Raemma p Luck, MD, Principal Investigator — Temple University
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Al-Qattan MM. Vicryl Rapide versus Vicryl suture in skin closure of the hand in children: a randomized prospective study. J Hand Surg Br. 2005 Feb;30(1):90-1. doi: 10.1016/j.jhsb.2004.08.005. PMID 15620501
- [Derived] Tejani C, Sivitz AB, Rosen MD, Nakanishi AK, Flood RG, Clott MA, Saccone PG, Luck RP. A comparison of cosmetic outcomes of lacerations on the extremities and trunk using absorbable versus nonabsorbable sutures. Acad Emerg Med. 2014 Jun;21(6):637-43. doi: 10.1111/acem.12387. PMID 25039547
- See also: abstract of Vicryl Rapide and RCT — http://www.ncbi.nlm.nih.gov/sites/entrez
- See also: use of absorbable sutures in pediatric facial lacerations — http://emergency-medicine.jwatch.org/cgi/content/full/2008/425/1
- See also: review of wound management, sutures — http://emedicine.medscape.com/article/884838-overview